CLINICAL TRIAL: NCT03565653
Title: The Effects of Dietary Salt on Post-exercise Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1085139
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Blood Pressure; Post-Exercise Hypotension
MeSH Terms: conditions — Post-Exercise Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dietary salt (Experimental): For 10 days each, participants will be asked to eat a recommended sodium diets (2300 mg Na+/d) while taking unmarked pills containing uniodized table salt. On the 10th day, participants will report to the lab to complete 60 minutes of cycling exercise. Following exercise, participants will rest for 60 minutes while undergoing serial blood pressure measurements. Participants will then be outfitted with ambulatory blood pressure cuffs for assessment of blood pressure over the following 24 hours.
  Interventions: Other: High dietary salt
- Placebo (Experimental): For 10 days each, participants will be asked to eat a recommended sodium diets (2300 mg Na+/d) while taking unmarked pills containing a placebo (dextrose). Participants will complete both interventions in random order. On the 10th day, participants will report to the lab to complete 60 minutes of cycling exercise. Following exercise, participants will rest for 60 minutes while undergoing serial blood pressure measurements. Participants will then be outfitted with ambulatory blood pressure cuffs for assessment of blood pressure over the following 24 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: High dietary salt — ~4,000 mg Na+/day
  Arms: High dietary salt
Other: Placebo — dextrose
  Arms: Placebo

SUMMARY:
The new American Heart Association (AHA) blood pressure guidelines are expected to raise the prevalence of high blood pressure to ~46% in the United States. One recommendation for lowering blood pressure is aerobic exercise, which produces a period of lowered blood pressure (post-exercise hypotension; PEH) that lasts up to 24 hours. It is believed that PEH may be responsible for the observations of lowered blood pressure following initiation of exercise. However, most Americans eat too much salt, which expands plasma volume and may prevent PEH, rending aerobic exercise ineffective in improving blood pressure status.

DETAILED DESCRIPTION:
Recently released blood pressure guidelines from the American Heart Association and American College of Cardiology are expected to raise the prevalence of hypertension in America from ~33% to ~46%. A single bout of aerobic exercise produces a prolonged period (up to 24 hours) of lowered blood pressure (post-exercise hypotension; PEH). Repeated bouts of aerobic exercise results in maintenance of lowered blood pressure, leading to recommendations of aerobic exercise for improvement of blood pressure status. However, more than 90% of Americans consume more sodium in their diets than is recommended. This is alarming, as excess dietary sodium intake expands plasma fluid volume, which may in turn attenuate the reduction in BP following exercise. Therefore, the objective of this project is to determine the effects of high dietary sodium intake on PEH. The investigators hypothesize that, compared to a recommended sodium diet, a high salt diet will attenuate post-exercise hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active

Exclusion Criteria:

* high blood pressure (>140/90 mmHg)
* history of cardiovascular disease
* history of cancer
* history of diabetes
* history of kidney disease
* obesity (BMI > 30 kg/m2)
* smoking or tobacco use
* current pregnancy
* nursing mothers
* communication barriers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Post-exercise hypotension | 24 hours following exercise
  Change in mean arterial pressure from pre- to post-exercise

SECONDARY OUTCOMES:
Blood pressure reactivity | 10th day of high salt diet
  Change in mean, systolic, and diastolic blood pressure from baseline to exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No